CLINICAL TRIAL: NCT03936270
Title: Palbociclib Plus Letrozole Treatment After Progression to Second Line Chemotherapy for Women With ER/PR-positive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 1018
Record Dates: First submitted 2019-02-05; First posted 2019-05-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
Keywords: Palbociclib; Letrozole; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib 125mg + Letrozole 2.5mg (Experimental): Palbociclib 125mg per day, administered orally in 4-week cycles (3 weeks of treatment followed by 1 week off) PLUS Letrozole 2.5mg per day administered orally (continuous treatment).
  Interventions: Drug: Palbociclib 125mg; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Palbociclib 125mg — The Palbociclib capsules supplied for this study contains 75 mg, 100 mg or 125 mg of Palbociclib. It must be taken orally 125 mg once daily for 21 consecutive days followed by 7 days off treatment (Schedule 3/1) to comprise a complete cycle of 28 days.
  Other Names: Ibrance®
Drug: Letrozole 2.5mg — Letrozole will be supplied as a 2.5 mg film-coated tablet. It must be taken at the recommended dose of 2.5 mg once daily.
  Other Names: Femara

SUMMARY:
The primary objective of this study is to evaluate 12 weeks progression-free survival (PFS) rate of Palbociclib plus Letrozole in ER/PR positive endometrioid or high-grade serous ovarian cancer who have disease progression on second-line chemotherapy.

DETAILED DESCRIPTION:
Letrozole (Femara®) is an oral non-steroidal aromatase inhibitor that is approved worldwide for the treatment of postmenopausal women with breast cancer. It is administered orally on a continuous 2.5 mg daily dosing regimen and has a good toxicity profile. Palbociclib (Ibrance®) is an active potent and highly selective reversible inhibitor of cyclin- dependent kinases 4 and 6 (CDK4/6). Palbociclib was approved by the United States Food and Drug Administration (U.S. FDA) and the European Medicines Agency (EMA) for the treatment of postmenopausal women with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced or metastatic breast cancer in combination with an aromatase inhibitor based on a randomized, double-blind, placebo-controlled, international clinical trial PALOMA-2. It is administered orally on a dose of 125 mg per day in 4-week cycles (3 weeks of treatment followed by 1 week off). This trial was based on preclinical studies that showed a synergistic effect between targeting the ER and cyclin-D-CDK4/6-Rb pathway. The principal toxicity was myelotoxicity but it was managed with appropriate supportive care and dose reductions13.

Based on the results of phase 1 and 2 clinical trials of CDK4/6 inhibitors used as monotherapy to treat patients with recurrent ovarian cancer, we hypothesized that, as Palbociclibe is active in this population and many ovarian cancer show ER/PR expression, its combination with Letrozole can improve outcomes in ER/PR positive endometrioid or high-grade serous Ovarian Cancer who have disease progression on second-line chemotherapy, similar to what is seen in breast cancer studies.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study;
2. Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
3. 18 years of age or older;
4. Patient agrees not to participate in another interventional study while on treatment;
5. Histology confirmed ovarian cancer serous or endometrioid high degree, fallopian tube or with locoregional recurrence peritoneum (not amenable to curative treatment) or metastatic;
6. Estrogen (ER) and/or progesterone (RP) receptor positive tumor, defined as > 10% by immunohistochemical examination in the local laboratory;
7. Availability of tumor sample from the primary tumor or metastasis, fixed in formalin and embedded in paraffin, for confirmation of positivity for ER and/or RP in a central laboratory;
8. Disease measurable by RECIST 1.1 as assessed by the local investigator or radiologist;
9. Patients must have chemotherapy application for recurrence locoregional or metastatic according to the following criteria:

   * at least one platinum-based chemotherapy regimen;
   * have confirmed no more than 3 chemotherapy regimens for locally advanced or metastatic disease
10. Patient must have radiographic disease progression to last treatment;
11. Functional capacity by the Eastern Cooperative Oncology Group (ECOG) ≤ 2;
12. Adequate bone marrow function:

    * Absolute neutrophil count (CAN) ≥ 1,500/mm3 (≥ 1.5x109/L)
    * Plates ≥ 100,000/mm3 or ≥ 100 x 109/L
    * Hemoglobin ≥ 9.0 g/dL;

12. Adequate liver function:

* Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤ 3.0 x ULN if there is Gilbert's Syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN (≤ 5.0 x ULN if liver tumor was involved)
* Alkaline phosphatase ≤ 2.5 x ULN (≤ 5.0 x ULN if any liver tumor involvement); 13. Adequate kidney function:
* Estimated creatinine clearance ≥ 15 mL/min; 14. Evidence of lack of potential to become pregnant:
* Post-menopause (defined as at least 1 year without menstruation) before selection, or
* Radiotherapy-induced oophorectomy with the last menstruation > 1 year ago, or
* Surgical sterilization (bilateral oophorectomy or hysterectomy).

Exclusion Criteria:

1. Patients with a known hypersensitivity to Palbociclib or Letrozole or any of the excipients of the product;
2. Previous treatment with CDK4/6 inhibitors or endocrine therapy;
3. Disease progression during or within 6 months of the first platinum-based chemotherapy regimen.
4. Persistent toxicities (Grade 2 or higher) caused by previous anticancer therapy (excluding alopecia);
5. Patients with a second primary cancer, except: adequately treated non-melanoma skin cancer, cervical cancer in situ curatively treated, Ductal carcinoma in situ (DCIS), stage 1 grade 1 endometrial carcinoma curatively treated with no evidence of illness for 3 years;
6. Last dose of chemotherapy or radiotherapy within 3 weeks of study enrollment;
7. Patients with symptomatic uncontrolled brain metastases. An exam to confirm the absence of brain metastases is not necessary;
8. Major surgical procedure within 3 weeks prior to study randomization, or planned during the course of the study;
9. Patients considered a precarious medical risk due to a disorder uncontrolled serious medical, non-malignant systemic disease, or uncontrolled active infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent myocardial infarction (within 6 months), stroke, gastrointestinal bleeding, or any psychiatric disorder that precludes informed consent;
10. Patients who have difficulty taking oral medication or any digestive tract dysfunction or inflammatory bowel disease that interferes with intestinal absorption of medications (eg, partial bowel obstruction or malabsorption);
11. Patients received potent inhibitors or inducers of CYP3A4 within 7 days of randomization;
12. Pregnant or nursing women;
13. The patient has a known history of testing positive for human immunodeficiency virus (HIV);
14. Patients with known liver disease (ie, Hepatitis B or C);
15. Treatment with any product under investigation during the last 28 days;
16. Other acute or chronic medical or psychiatric condition or severe laboratory abnormality that could increase the risk associated with participation in the study or that could interfere with the interpretation of the study results and, in the investigator's judgment, would make the research participant unsuitable for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Twelve weeks of Progression Free Survival | 12 weeks
  The primary objective of this study is to evaluate 12 weeks progression-free survival (PFS) rate of Palbociclib plus Letrozole in ER/PR positive endometrioid or high-grade serous ovarian cancer who have disease progression on second-line chemotherapy.

SECONDARY OUTCOMES:
Overall response | 2 years
  defined as the proportion of patients who have a partial or complete response to therapy according to RECIST 1.1
Overall Survival | 2 years
  Overall Survival at year 1 and 2
Clinical Benefit Rate | 2 years
  defined as the proportion of patients who have achieved complete response, partial response and stable disease for at least 24 weeks.
Duration of response | 2 years
  defined as the time from response to progression by RECIST v11.1 or death
CA-125 response (GCIG criteria) | 2 years
  defined as the proportion of patients who have achieved at least a 50% reduction in CA 125 levels from a pretreatment sample (must be confirmed and maintained for at least 28 days)
Time to progression by CA-125 (GCIG criteria) or RECIST | 2 years
  defined as the time from response to progression by CA 125 (GCIG criteria) or RECIST
Quality of Life (FACT-O questionnaire) | 2 years
  assessed using the FACT-O questionnaire
Safety (adverse events) | 2 years
  defined as the proportion of patients who present adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Bronzon Damian, Principal Investigator — Latin American Cooperative Oncology Group
Locations (5):
- Brazil (5):
  - UFMG - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No